CLINICAL TRIAL: NCT07281937
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2b Study of Weekly Oral Ecnoglutide (VRB-101) in Participants Who Have Obesity or Overweight With Weight-Related Comorbidities
Brief Title: A Study of Weekly Oral Ecnoglutide (VRB-101) in Participants Who Have Obesity or Overweight With Weight-Related Comorbidities
Acronym: EVOLVE-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Verdiva Bio Dev Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VRB-101-201
Record Dates: First submitted 2025-12-04; First posted 2025-12-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
Keywords: Hypertension; Weight reduction; Dose Escalation; Glucagon-like peptide-1 (GLP-1)
MeSH Terms: conditions — Obesity; Overweight; Hypertension; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Schedule A: VRB-101 (Active Arm 1) (Experimental): Participants will receive VRB-101 once every week.
  Interventions: Drug: VRB-101
- Schedule A: VRB-101 (Active Arm 2) (Experimental): Participants will receive VRB-101 once every week.
  Interventions: Drug: VRB-101
- Schedule A: VRB-101 (Active Arm 3) (Experimental): Participants will receive VRB-101 once every week.
  Interventions: Drug: VRB-101
- Schedule B: VRB-101 (Active Arm 4) (Experimental): Participants will receive VRB-101 once every week.
  Interventions: Drug: VRB-101
- Schedule B: VRB-101 (Active Arm 5) (Experimental): Participants will receive VRB-101 once every week.
  Interventions: Drug: VRB-101
- Pooled Placebo (Placebo Comparator): Participants will receive matching placebo to VRB-101 once every week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VRB-101 — VRB-101 tablets will be administered orally.
  Other Names: Oral Ecnoglutide
  Arms: Schedule A: VRB-101 (Active Arm 1); Schedule A: VRB-101 (Active Arm 2); Schedule A: VRB-101 (Active Arm 3); Schedule B: VRB-101 (Active Arm 4); Schedule B: VRB-101 (Active Arm 5)
Drug: Placebo — Placebo tablets will be administered orally.
  Arms: Pooled Placebo

SUMMARY:
The aim of this study is to evaluate the efficacy of VRB-101 for body weight reduction compared to placebo in participants who have obesity or overweight with weight-related comorbidities.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study of oral ecnoglutide (VRB-101), with 5 active arms and 1 placebo arm. The study will include a Screening Period of 4 weeks, followed by a 20-week Study Treatment Period and a 4-week Safety Follow-up Period prior to the end of study (EOS) visit.

ELIGIBILITY:
Inclusion Criteria:

* Have hemoglobin A1c (HbA1c) <6.5%.
* Have a BMI of ≥30 kg/m2 OR ≥27 kg/m2 and <30 kg/m2 with at least 1 weight-related comorbidity.
* Have a self-reported history of stable body weight for the 3 months prior to randomization (≤5% body weight change).
* Participants of childbearing potential must be non-pregnant and non-lactating and must agree to use study-specified contraceptive methods.

Exclusion Criteria:

* Have any prior diagnosis of type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM), or other forms of diabetes mellitus. A participant with a history of gestational diabetes may be included in the study if the participant has an HbA1c < 6.5% at Screening.
* Have at least 1 laboratory value suggestive of diabetes during Screening, including 1 or more of HbA1c ≥6.5% (48 mmol/mol) or random glucose ≥200 mg/dL (11.1 mmol/L).
* Have had exposure to glucagon-like peptide -1 (GLP-1) 6 months prior to Screening or any prior history of known or suspected hypersensitivity/allergies, intolerability, or lack of efficacy to these medications. Have known or suspected hypersensitivity to study intervention(s), to selective GLP-1 receptor agonist (RA) or glucose-dependent insulinotropic peptide (GIP)/GLP-1 or GLP-1/glucagon (GCG) dual receptor agonists.
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time within the dosing period, including follow -up, and for at least 60 days after the last dose of study intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mean percent change from baseline in body weight | From Baseline (Day 0) up to Week 21
  To evaluate the efficacy of VRB-101 for body weight reduction compared to placebo in Schedule A dose regimens.

SECONDARY OUTCOMES:
Absolute change from baseline in body weight | From Baseline (Day 0) up to Week 21
  To compare the effect of VRB-101 versus placebo on body weight in Schedule A.
Percentage of participants who achieve 5% or more body weight reduction | From Baseline (Day 0) up to Week 21
  To compare the effect of VRB-101 versus placebo on body weight in Schedule A
Change from baseline in body mass index (BMI) | From Baseline (Day 0) up to Week 21
  To compare the effect of VRB-101 versus placebo on body weight in Schedule A.
Number of study participants with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | From Baseline (Day 0) up to Week 24
  To assess safety and tolerability of study interventions. Adverse events (AEs) reported after first administration of study intervention will be designated as a TEAE.
Change from baseline in blood pressure (BP) | From Baseline (Day 0) up to Week 24
  To assess safety and tolerability of study interventions.
Change from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | From Baseline (Day 0) up to Week 21
  To assess safety and tolerability of study interventions.
  C-SSRS is a tool to help systematically assess suicidal ideation and behavior in participants during clinical studies of centrally acting drugs. It is composed of 3 questions addressing suicidal behavior and 5 questions addressing suicidal ideation, with sub-questions assessing the severity. The responses to the questions will be recorded as 'yes/no'.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Clinical Study Site 103, Anniston, Alabama
  - Clinical Study Site 109, Cullman, Alabama
  - Clinical Study Site 110, Phoenix, Arizona
  - Clinical Study Site 113, Little Rock, Arkansas
  - Clinical Study Site 111, Anaheim, California
  - Clinical Study Site 107, Montclair, California
  - Clinical Study Site 118, Tarzana, California
  - Clinical Study Site 119, Decatur, Georgia
  - Clinical Study Site 116, West Des Moines, Iowa
  - Clinical Study Site 106, Wichita, Kansas
  - Clinical Study Site 122, Southfield, Michigan
  - Clinical Study Site 121, Omaha, Nebraska
  - Clinical Study Site 117, Binghamton, New York
  - Clinical Study Site 101, Rochester, New York
  - Clinical Study Site 120, Charlotte, North Carolina
  - Clinical Study Site 108, Monroe, North Carolina
  - Clinical Study Site 105, Norman, Oklahoma
  - Clinical Study Site 114, Duncansville, Pennsylvania
  - Clinical Study Site 115, Knoxville, Tennessee
  - Clinical Study Site 112, Dallas, Texas
  - Clinical Study Site 102, San Antonio, Texas
  - Clinical Study Site 104, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No